CLINICAL TRIAL: NCT02619058
Title: An Open Label, Dose Escalation, Phase I Clinical Trial of Adoptive Transfer With Autologous NKT Cells in Metastatic Melanoma Patients
Brief Title: A Clinical Trial of Adoptive Transfer With Autologous NKT Cells in Metastatic Melanoma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCH-MM-150620
Record Dates: First submitted 2015-11-19; First posted 2015-12-02 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma
Keywords: NKT; metastatic melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1（NKT cells single low dose） (Experimental): Patients will receive intravenous administration of autologous NKT cells, the dose level is 1×10^9 on d1, 2×10^9 on d3, 4×10^9 on d29, 8×10^9 on d31.
  Interventions: Biological: NKT cells
- Arm 2（NKT cells single high dose） (Experimental): Patients will receive intravenous administration of autologous NKT cells, the dose level is 5×10^9 on d1, 5×10^9 on d3, 5×10^9 on d29, 5×10^9 on d31.
  Interventions: Biological: NKT cells
- Arm 3（NKT cells multiple dose） (Experimental): Patients will receive intravenous administration of autologous NKT cells, the dose level is 5×10^9 on d1, 5×10^9 on d3 of each 28 days-cycle, the dosing will be ended after 8 cycles.
  Interventions: Biological: NKT cells

INTERVENTIONS:
Biological: NKT cells — autologous natural killer T cell

SUMMARY:
Considerable progress in the treatment of metastatic melanoma has been made in the past 5years, with the approval of immune checkpoint-blocking antibodies and agents targeting BRAF mutation. Investigators conducted a open label, dose escalation, phase I clinical trial of to explore the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of intravenous administration of autologous NKT Cells in metastatic melanoma patients.

DETAILED DESCRIPTION:
Considerable progress in the immunotherapy of metastatic melanoma has been made in the past 5 years, with the approval of immune checkpoint-blocking antibodies. NKT cells are a potent immunoregulatory cell population heavily implicated in promoting immunity to infection and cancer. And now with new generation of amplification method, more than 1,000 folds amplification of NKT cells can be obtained, so NKT cell based adoptive cell transfer is now available and might show its efficacy in melanoma. Investigators conducted this open label, dose escalation, phase I clinical trial of to explore the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of intravenous administration of autologous NKT Cells in metastatic melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathological or cytologically confirmed malignant melanoma with unresectable Stage III or Stage IV (including skin and distant lymph node metastasis M1a, lung metastasis M1b).
* Patients who are resistant /refractory to approved therapies, or for whom no curative therapies are available.
* Male or female, aged ≥18 and ≤70 years; ECOG performance status score of 0-2; Life expectancy of at least six months.
* For women of childbearing potential, a negative pregnancy test within 7 days prior to the first treatment.
* At least four weeks since prior other anti-tumor therapy, including endocrine, chemotherapy/radiotherapy and targeted therapy, at least six weeks since prior nitrosourea and mitomycin dosing, and have recovered from the adverse reactions due to prior therapy.
* At least 4 weeks before prior surgery.
* Must have one measurable or evaluable lesion according to RECIST 1.1
* With enough tumor tissues and diagnosed by the designated laboratory.
* Body weight >50kg.
* Without functional disorder of major organs ( laboratory examination): Neutrophils≥1.5×10^9/L, lymphocyte≥1.0×10^9/L, PLT≥100×10^9/L, Hb≥110g/L; BUN and Cr within normal range; TBIL≤1.5 times upper limit; ALT/AST≤2.5 times upper limit; PT/APTT within normal range.
* Without obvious hereditary disease.
* Must sign a written informed consent form prior to entering the study, with good compliance.

Exclusion Criteria:

* With extrapulmonary metastatic of melanoma, for instance, distant metastasis of liver, brain, bone, adrenal gland.
* With serious internal disease, including serious heart disease, cerebral vascular disease, uncontrolled diabetes, uncontrolled hypertension, serious infections, active peptic ulcer, renal failure and respiratory failure.
* Uncontrolled infectious diseases or other serious diseases, for example, HIV, Hepatitis B and Hepatitis C.
* Uncontrolled brain metastases.
* Lymphoma or leukemia patients.
* Patients who have received bone marrow, stem cells or organ transplantation.
* With immunodeficiency or autoimmune disease, leucoderma excluded.
* Allergic constitution.
* Chronic diseases needed immunosuppressive therapy or hormone therapy.
* Patients treated with steroid hormone.
* Unable to evaluate the immune status, or patients cannot comply with follow-up clinical evaluation.
* Patients diagnosed with MDS (myelodysplastic syndromes).
* Patients who are pregnant or breast-feeding.
* Women (or patients' wife) of child-bearing without effective contraceptive measures.
* Patients receiving any investigational drug or investigational treatment within 4 weeks prior to first dosing.
* With uncontrolled mental disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experiencing at least one dose limiting toxicity (DLT) of intravenous administration of autologous NKT Cells in metastatic melanoma patients. | 252 days
  DLT is defined as any of the following toxicities assessed as at least possibly related to NKT cells by the investigator up to 28 days each cycle(up to 8 cycles,with 28 days' safety and efficacy follow-up after the end of the last cycle) after the end of adoptive transfer: any Grade greater than or equal to (>=) 3 non-hematological toxicity, but excluding the conditions mentioned in the protocol; any Grade 4 neutropenia of greater than (>)5 days duration or Grade >=3 febrile neutropenia; any Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding; any Grade 4 anemia.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD,PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Hoos A, Parmiani G, Hege K, Sznol M, Loibner H, Eggermont A, Urba W, Blumenstein B, Sacks N, Keilholz U, Nichol G; Cancer Vaccine Clinical Trial Working Group. A clinical development paradigm for cancer vaccines and related biologics. J Immunother. 2007 Jan;30(1):1-15. doi: 10.1097/01.cji.0000211341.88835.ae. PMID 17198079
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295